CLINICAL TRIAL: NCT07002411
Title: Hospitality Oriented Service Perception Evolution With Robots (HOSPER)
Acronym: HOSPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INRCA_008_2024
Record Dates: First submitted 2025-05-14; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Quality of Hospital Entrance Reception; Social Robots
Keywords: Older people

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM 1 (Experimental): Older subjects attending the INRCA hospital entrance
  Interventions: Other: Innovative hospital reception service with social robot NAO
- ARM 2 (Active Comparator): Older subjects attending the INRCA hospital entrance
  Interventions: Other: Innovative hospital reception service with social robot PEPPER

INTERVENTIONS:
Other: Innovative hospital reception service with social robot NAO — The robot NAO welcomes the user and asks how it can assist them. At this point, the user responds, and the robot, in turn, replies in two possible ways: If it has not understood the request, it prompts the user to rephrase it, and the process returns to the previous point. If it has understood the request, it explains the route the user needs to follow. Once the interaction has been successful or two consecutive attempts have failed, the robot asks the user if the necessary information has been provided. If yes, the robot dismisses the user. If no, the interaction resumes from the point where the robot asks for the department to reach or the exam to take.
  Arms: ARM 1
Other: Innovative hospital reception service with social robot PEPPER — The robot PEPPER welcomes the user and asks how it can assist them, stating the following phrase: "Good morning and welcome to INRCA. I am PEPPER and I am here to provide directions to help you reach your desired location within the hospital. Which department do you need to reach or which exam do you need to take? " At this point, the user responds, and the robot, in turn, replies in two possible ways: If it has not understood the request, it prompts the user to rephrase it, and the process returns to the previous point. If it has understood the request, it explains the route the user needs to follow. Once the interaction has been successful or two consecutive attempts have failed, the robot asks the user if the necessary information has been provided. If yes, the robot dismisses the user as follows: "Thank you for your participation. Have a good day." If no, the interaction resumes from the point where the robot asks for the department to reach or the exam to take.
  Arms: ARM 2

SUMMARY:
The HOSPER project aims to determine if using Pepper and NAO social robots at the IRCCS INRCA in Ancona's (Italy) entrance is a viable way to improve the current reception and guidance services for hospital visitors. The robots will offer proactive assistance and directions to departments.

DETAILED DESCRIPTION:
The primary aim of the "HOSPER" project is to assess the feasibility of an innovative reception and proactive guidance service designed to enhance the quality of the existing service provided by the IRCCS INRCA in Ancona (Italy). This will be achieved through the deployment of two social robots, Pepper and NAO, located at the hospital entrance to provide information to users inquiring about directions to specific departments. Furthermore, the study will evaluate the level of participant satisfaction with their interactions with the robots.

ELIGIBILITY:
Inclusion Criteria:

* Possession of full cognitive capacity;

Exclusion Criteria:

* • Lack of written informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
perceived quality of the innovative reception service | immediately after the intervention
  The perceived quality will be evaluated by an ad hoc Customer Satisfaction questionnaire. The definition of this indicator is evaluated by quantifying several variables, including: the attention received from the robot in terms of accuracy of the interaction and courtesy (score from 1 - not at all satisfied - to 7 - very satisfied), the clarity and completeness of the information received (score from 1 - not at all satisfied - to 7 - very satisfied), the respect for personal privacy (score from 1 - not at all satisfied - to 7 - very satisfied), the overall satisfaction with the service provided (score from 1 - not at all satisfied - to 7 - very satisfied), and whether the service would be recommended to others (score from 1 - absolutely not - to 7 - definitely yes).

SECONDARY OUTCOMES:
Usability | immediately after the intervention
  The usability will be evaluated by the System Usability Scale (SUS). It consists of a 10-item questionnaire with five response options for respondents, ranging from "Strongly Agree" to "Strongly Disagree." The score for the System Usability Scale (SUS) is calculated by following these steps:
  * For odd-numbered questions (1, 3, 5, 7, 9), subtract 1 from the user's rating.
  * For even-numbered questions (2, 4, 6, 8, 10), subtract the user's rating from 5.
  * Add the new values for all 10 questions.
  * Multiply this sum by 2.5. This final number gives you a score out of 100.
  The System Usability Scale (SUS) score, ranging from 0 to 100, is interpreted to indicate the perceived usability of a system. Higher scores suggest better usability.
  Interpreting SUS Scores:
  90-100: exceptionally good usability. 80-89: very good usability 70-79: good usability 60-69: the usability is marginal 50-59: Poor usability 0-49: Extremely poor usability

CONTACTS AND LOCATIONS:
Overall Officials: Letizia Ferrara, MD, Principal Investigator — IRCCS INRCA, Ancona, Italy
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No